CLINICAL TRIAL: NCT02023294
Title: Prospective Randomized Clinical Trial Comparing COnventional Laparoscopic Sleeve Gastrectomy Versus Endograb-assisted Single-port Sleeve Gastrectomy
Brief Title: Conventional Laparoscopic Sleeve Gastrectomy Versus Endograb-assisted Single-port Sleeve Gastrectomy
Acronym: GTLEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Salvador Morales Conde, Innovation and Minimally Invasive Surgery Unit Cordinator, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTL-EG-01
Record Dates: First submitted 2013-12-10; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lap (Active Comparator): Patients candidate to bariatric surgery undergoing Conventional laparoscopic Sleeve Gastrectomy
  Interventions: Procedure: Convetional laparoscopic Sleeve Gastrectomy
- SILS (Experimental): Patients candidate to bariatric surgery undergoing Single Incision Laparoscopic Sleeve Gastrectomy supported by Endograb
  Interventions: Procedure: SILS Sleeve gastrectomy

INTERVENTIONS:
Procedure: Convetional laparoscopic Sleeve Gastrectomy — Convetional laparoscopic sleeve gastrectomy using 5 ports (incisions) in the abdominal wall
  Arms: Lap
Procedure: SILS Sleeve gastrectomy — Single incision Sleeve gastrectomy using only one port (incision) on the abdominal wall assisted by an special Traction Device for single port surgery (Endograb)
  Other Names: Endograb™ (Virtual Ports, Misgav, Israel)
  Arms: SILS

SUMMARY:
Bariatric surgery has been established as the best treatment for morbid obesity, compared with diet or medical treatment. Laparoscopic approach have improved the results of this surgery in terms of postoperative pain, reduction in the number of complications and hospital stay, as well as better cosmetic results. Conventional laparoscopic technique requires five to seven abdominal incisions to facilitate placement of the multiple trocars. New Single Incision Laparoscopic Surgery (SILS)has been developed as a new technique where only one incision is needed for the introduction of all trocars. Altough this technique can be performed with conventional laparoscopic instruments, new devides have been developed for facilitate this operations by SILS. The investigators think that reducing the number of incision would decrease the postoperative pain and improve cosmetic results in our patients, being a safe and technically feasible intervention supported by these special devices.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index > 40
* Body Mass Index > 35 with 2 mayor comorbidities

Exclusion Criteria:

* Severe gastroesophageal reflux
* Esophagitis grade B or higher
* Midline periumbilical incision
* Umbilical hernia >4cms.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 3 days
  Postoperative pain is assessed using a visual analog scale (VAS)on the first 3 postoperative days

SECONDARY OUTCOMES:
Cosmestic results | 1,3 and 6 months
  Cosmetic results will be assess using visual analog scale (VAS)at 1,3 and 6 months after surgery
Operative time | Surgery
  operative time will be compared between two thechniques

OTHER OUTCOMES:
Perioperative complications | 1 month
  Appearence of intraoperative and postoperative complications derived from the technique will be recorded an compared with the two techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Morales Conde Salvador, phD, Principal Investigator — Hospital Universitario Virgen del Rocio; Alarcón del Agua Isaías, PhD, Study Chair — Hospital Universitario Virgen del Rocio
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Seville, Spain

REFERENCES:
- [Background] Morales-Conde S, Garcia Moreno J, Canete Gomez J, Barranco Moreno A, Socas Macias M. [Single incision laparoscopic right hemicolectomy due to cancer of the colon]. Cir Esp. 2010 Aug;88(2):129-31. doi: 10.1016/j.ciresp.2009.07.016. Epub 2009 Oct 31. No abstract available. Spanish. PMID 19880099
- [Background] Martin-Cartes J, Morales-Conde S, Suarez-Grau J, Lopez-Bernal F, Bustos-Jimenez M, Cadet-Dussort H, Socas-Macias M, Alamo-Martinez J, Tutosaus-Gomez JD, Morales-Mendez S. Use of hyaluronidase cream to prevent peritoneal adhesions in laparoscopic ventral hernia repair by means of intraperitoneal mesh fixation using spiral tacks. Surg Endosc. 2008 Mar;22(3):631-4. doi: 10.1007/s00464-007-9423-5. PMID 17593452
- [Background] Feliu-Pala X, Martin-Gomez M, Morales-Conde S, Fernandez-Sallent E. The impact of the surgeon's experience on the results of laparoscopic hernia repair. Surg Endosc. 2001 Dec;15(12):1467-70. doi: 10.1007/s00464-001-9017-6. PMID 11965467